CLINICAL TRIAL: NCT01690338
Title: A Perspective, Multicentre, Randomized，Blind Study of Residual Curarization Incidence in China
Brief Title: A Study of Residual Curarization Incidence in China
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Ruijin Hospital (Other); RenJi Hospital (Other); Shanghai Zhongshan Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); West China Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Zhujiang Hospital (Other); Chinese PLA General Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Tianjin Medical University General Hospital (Other); Xiangya Hospital of Central South University (Other); Central South University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Peking Union Medical College Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); China Medical University Hospital (Other); Hebei Medical University Fourth Hospital (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Xinmin Wu, Clinical Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSA-NMB-001
Record Dates: First submitted 2012-09-04; First posted 2012-09-21 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Perioperative/Postoperative Complications; PORC (Postoperative Residual Curarization)
Keywords: TOFr (train of four ratio); airway extubation; PACU (postanesthesia care unit); PORC (postoperative residual curarization)
MeSH Terms: conditions — Postoperative Complications; Delayed Emergence from Anesthesia | interventions — Vecuronium Bromide; Rocuronium; cisatracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vecuronium Bromide (Active Comparator): Patients who will be performed general anesthesia and tracheal intubation. Vecuronium will be used during surgery and tracheal extubation is scheduled when surgery is over.
  Interventions: Drug: Vecuronium Bromide
- cisatracurium (Active Comparator): Patients who will be performed general anesthesia and tracheal intubation. Cisatracurium will be used during surgery and tracheal extubation is scheduled when surgery is over.
  Interventions: Drug: Cisatracurium
- rocuronium (Active Comparator): Patients who will be performed general anesthesia and tracheal intubation. Rocuronium will be used during surgery and tracheal extubation is scheduled when surgery is over.
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Vecuronium Bromide — Administrative protocol of Vecuronium Bromide is determined by each caregiver's clinical experience.
  Other Names: Norcuron
  Arms: Vecuronium Bromide
Drug: Rocuronium — Administrative protocol of rocuronium is determined by each caregiver's clinical experience.
  Other Names: Esmeron
  Arms: rocuronium
Drug: Cisatracurium — Administrative protocol of cisatracurium is determined by each caregiver's clinical experience
  Other Names: Nimbex
  Arms: cisatracurium

SUMMARY:
The purpose of this study is to determine the incidence of residual curarization in PACU and relevant risk factors.

DETAILED DESCRIPTION:
In the last twenty years, residual curarization in PACU (Post Anesthesia Care Unit) has become a common problem in clinical practice and poses high risk to patients. The residual curarization incidence of Neuromuscular blocking agents (NMBA) varies very much between different studies. These differences indicates the necessity of further study. In China, there is no common view of the harmfulness of residual curarization and its complications. The consensus on the necessity of neuromuscular transmission monitoring and neuromuscular blockade antagonist has not been reached yet. There is also no similar large-scale survey in China. In this case, the investigators conduct this large scale multicentre study, which is designed to learn the incidence of residual curarization and its complications. Further analysis of risk factors will also been made. All these efforts are hoped to fill the data gap and provide reliable evidences for rational use of NMBA.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Nondepolarized NMBA will be given during surgery and tracheal extubation will be performed after surgery
* Willing to comply with all study procedures and provide signed and dated informed consent

Exclusion Criteria:

* Allergic reaction to gel electrode
* Neuromuscular disorders and hepatic or renal dysfunction
* Scheduled to receive mechanical ventilation therapy
* Involved in other clinical trials
* Body position and surgical procedure affecting TOF-Watch SX normal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6090 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
incidence of TOFr<0.9 | From tracheal extubation to 1 minute after extubation
  Once tracheal extubation is performed after the surgery is over, monitor the neuromuscular transmission function (TOF ratio) immediately.

SECONDARY OUTCOMES:
Incidence of TOFr<0.9 | One minute after arriving at PACU
  When patients arrive at PACU(an expected average of 15 minutes after surgery is over), monitor the neuromuscular transmission function (TOF ratio) immediately
Incidence of TOFr<0.7 | From tracheal extubation to 1 minute after extubation
  Once tracheal extubation is performed after the surgery is over, monitor the neuromuscular transmission function (TOF ratio) immediately.
Incidence of TOFr<0.7 | One minute after arriving at PACU
  When patients arrive at PACU(an expected average of 15 minutes after surgery is over), monitor the neuromuscular transmission function (TOF ratio) immediately

OTHER OUTCOMES:
any sign of residual curarization (listed in description below) | First 24h after surgery
  Sign of residual curarization :
  1. dyspnea
  2. weak hand-grip force
  3. Head lift or leg lift time shorter than 5s
  4. aspiration
  5. respiratory rate >20/min
  6. hypoxemia (SpO2<90% when O2>3L/min)
pulmonary complications (See description) | participants will be followed for the duration of hospital stay, an expected average of one week
  pulmonary complications
  1. pneumonia
  2. pulmonary atelectasis
  3. mechanical ventilation required

CONTACTS AND LOCATIONS:
Overall Officials: Xinmin Wu, Doctor, Principal Investigator — Peking University First Hospital
Locations (22):
- China (22):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital Southern Medical University, Guangzhou, Guangdong
  - Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Wuhan Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - China Medical University Hospital, Shenyang, Liaoning
  - Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality
  - RenJi Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital Of College of Medicine, Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Background] Cammu G, De Witte J, De Veylder J, Byttebier G, Vandeput D, Foubert L, Vandenbroucke G, Deloof T. Postoperative residual paralysis in outpatients versus inpatients. Anesth Analg. 2006 Feb;102(2):426-9. doi: 10.1213/01.ane.0000195543.61123.1f. PMID 16428537
- [Background] Naguib M, Kopman AF, Lien CA, Hunter JM, Lopez A, Brull SJ. A survey of current management of neuromuscular block in the United States and Europe. Anesth Analg. 2010 Jul;111(1):110-9. doi: 10.1213/ANE.0b013e3181c07428. Epub 2009 Nov 12. PMID 19910616
- [Background] Naguib M, Kopman AF, Ensor JE. Neuromuscular monitoring and postoperative residual curarisation: a meta-analysis. Br J Anaesth. 2007 Mar;98(3):302-16. doi: 10.1093/bja/ael386. PMID 17307778
- [Background] Hayes AH, Mirakhur RK, Breslin DS, Reid JE, McCourt KC. Postoperative residual block after intermediate-acting neuromuscular blocking drugs. Anaesthesia. 2001 Apr;56(4):312-8. doi: 10.1046/j.1365-2044.2001.01921.x. PMID 11284816
- [Background] Baillard C, Clec'h C, Catineau J, Salhi F, Gehan G, Cupa M, Samama CM. Postoperative residual neuromuscular block: a survey of management. Br J Anaesth. 2005 Nov;95(5):622-6. doi: 10.1093/bja/aei240. Epub 2005 Sep 23. PMID 16183681
- [Background] Cammu G, de Baerdemaeker L, den Blauwen N, de Mey JC, Struys M, Mortier E. Postoperative residual curarization with cisatracurium and rocuronium infusions. Eur J Anaesthesiol. 2002 Feb;19(2):129-34. doi: 10.1017/s0265021502000236. PMID 11999596
- [Background] Baillard C, Gehan G, Reboul-Marty J, Larmignat P, Samama CM, Cupa M. Residual curarization in the recovery room after vecuronium. Br J Anaesth. 2000 Mar;84(3):394-5. doi: 10.1093/oxfordjournals.bja.a013445. PMID 10793602
- [Background] Murphy GS, Szokol JW, Marymont JH, Franklin M, Avram MJ, Vender JS. Residual paralysis at the time of tracheal extubation. Anesth Analg. 2005 Jun;100(6):1840-1845. doi: 10.1213/01.ANE.0000151159.55655.CB. PMID 15920224
- [Background] Debaene B, Plaud B, Dilly MP, Donati F. Residual paralysis in the PACU after a single intubating dose of nondepolarizing muscle relaxant with an intermediate duration of action. Anesthesiology. 2003 May;98(5):1042-8. doi: 10.1097/00000542-200305000-00004. PMID 12717123
- [Background] Srivastava A, Hunter JM. Reversal of neuromuscular block. Br J Anaesth. 2009 Jul;103(1):115-29. doi: 10.1093/bja/aep093. Epub 2009 May 24. PMID 19468024